CLINICAL TRIAL: NCT07360574
Title: Piezo2-related Arthrogryposis & physiopathOLOgy 3
Acronym: PAOLO3
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0314
Record Dates: First submitted 2025-12-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arthrogryposis Multiplex Congenita; Piezo2 Mutation Gain of Function
Keywords: Arthrogyposis; Piezo2
MeSH Terms: conditions — Arthrogryposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days

SUMMARY:
Study type: Observational, non-interventional, single-center, descriptive study.

Goal of the study:

The goal of this observational study is to characterize the intensity, variability, and qualitative features of pain in patients with arthrogryposis multiplex congenita (AMC) caused by a gain-of-function mutation in PIEZO2. This population is rare and identified through the French national PARART registry (Pediatric and Adult Registry for patients with ARThrogryposis).

Population:

Participants are ≥10 years old, have a genetically confirmed gain-of-function PIEZO2 variant, and are registered in PARART. All procedures are conducted remotely; no onsite visit is required.

Main questions the study aims to answer:

* What is the intensity and day-to-day variability of pain over 14 consecutive days, measured with a Numerical Rating Scale (0-100)?
* What are the sensory qualities and anatomical distribution of pain in this population?
* How does this pain affect quality of life?
* What treatments (pharmacological or non-pharmacological) have been used, and how effective are they?

Study design:

There is no comparison group. The study is descriptive and aims to characterize the pain phenotype linked to PIEZO2 gain-of-function mutations.

What participants will do:

Participants will complete the following tasks remotely:

At Day 1:

Questionnaires:

* Saint-Antoine Pain Questionnaire (QDSA)
* SF-12
* EQ-5D-5L
* Pain monitoring: treatments used

For 14 consecutive days (Day 1 to Day 14), on a paper logbook:

* Daily self-reported Numerical Rating Scale (NRS, 0-100) for pain
* Daily body chart to document pain distribution

All data are collected through REDCap and a paper logbook. No clinical exam, biological sampling, or hospital visit is required.

The study duration for each participant is 14 days.

DETAILED DESCRIPTION:
Arthrogryposis multiplex congenita (AMC; Orpha code 1037) is a clinically and genetically heterogeneous group of disorders defined by congenital joint contractures affecting at least two distinct body regions (Dahan-Oliel et al. 2019).

Its estimated prevalence ranges from 1 in 3,000 to 1 in 12,000 live births, based on population-based epidemiological studies (Darin et al. 2002; Lowry et al. 2010; Hoff et al. 2012). The pathophysiology of AMC is closely linked to impaired fetal movement, with the severity of musculoskeletal manifestations depending on the timing and degree of fetal akinesia during development (Pollard, McGonnell, and Pitsillides 2014; Nowlan 2015; Felsenthal and Zelzer 2017).

Advances in molecular genetics have identified gain-of-function variants in the mechanosensitive ion channel PIEZO2 as a key etiology in a distinct subgroup of distal arthrogryposis (Coste et al. 2013). PIEZO2 plays a central role in mechanotransduction, converting mechanical stimuli into ionic currents in peripheral sensory neurons, thereby mediating proprioception and mechanical nociception (Wu, Lewis, and Grandl 2017; Szczot et al. 2021; Ma et al. 2023; Sánchez-Carranza et al. 2024).

Structural studies have shown that PIEZO2 forms a large trimeric propeller-shaped mechanosensitive channel whose architecture enables rapid transduction of membrane tension into cation influx, particularly Na⁺ and Ca²⁺ (Wang et al. 2019). Experimental data indicate that PIEZO2 gain-of-function mutations lead to delayed channel inactivation, neuronal hyperexcitability, and aberrant mechanotransduction, which likely underlie the distinctive pain phenotype observed in affected patients (Coste et al. 2013).

Clinically, individuals with PIEZO2-related AMC frequently report chronic diffuse pain with episodic exacerbations that are often poorly responsive to conventional analgesic strategies. Despite this recognizable pattern, genotype-phenotype correlations and the mechanisms driving pain severity and distribution remain insufficiently characterized.

This single-center, non-interventional observational study aims to describe the pain phenotype of individuals with AMC caused by gain-of-function variants in PIEZO2 identified through the national PARART registry (NCT05673265).

The study consists of prospective remote collection of self-reported outcomes using validated questionnaires. On Day 1, participants complete assessments of pain quality (QDSA) and quality of life (SF-12 and EQ-5D-5L), along with documentation of prior analgesic strategies. From Day 1 to Day 14, participants record daily pain intensity using a Numerical Rating Scale (0-100) and pain localization on a body chart, enabling evaluation of pain intensity, temporal variability, and anatomical distribution.

The study relies exclusively on descriptive statistical analyses, without hypothesis testing or comparison groups. Data are collected and managed using REDCap, in accordance with predefined procedures for pseudonymization, data integrity, and regulatory compliance (Harris et al. 2009; Harris et al. 2019). By systematically characterizing pain features and their impact on quality of life, this study seeks to improve understanding of the clinical pain profile associated with PIEZO2 gain-of-function mutations and to provide a foundation for future mechanism-based therapeutic strategies in this rare condition.

ELIGIBILITY:
Inclusion Criteria:

* PIEZO2 mutation gain of function
* Age ≥ 10 years
* Registered member of the PARART database (Pediatric and Adult Registry for Patients With ARThrogryposis)

Exclusion Criteria:

- Age < 10 years

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Arthrogryposis Multiplex Congenita with mutation gain of function of Piezo2 gene, followed by the University Hospital of Grenoble.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | From the start to the end of the follow-up at 14 days
  Quantitative Pain Evaluation : scale from 0 (no pain) to 100 (worst pain ever).

SECONDARY OUTCOMES:
Body Pain Map | From the start to the end of the follow-up at 14 days
  Location of the pain on the body.
EuroQol 5-Dimensions 5-Levels | At the start of the follow-up (Day 1).
  Self-questionnaire to evaluate the quality of life. 5D : Five Dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression).
  5L : Five Levels (No problems, Slight, Moderate, Severe, Extreme problems)
12-Item Short Form Health Survey | At the start of the follow-up (Day 1).
  The SF-12 is a self-reported questionnaire that produces two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Saint-Antoine Pain Questionnaire | At the start of the follow-up (Day 1).
  Qualitative description of pain with a variety of words refering to the different pain types, in distinct groups.
Pain Monitoring / Treatments | At the start of the follow-up (Day 1).
  Listing of pain treatments (medicinal or non-medicinal) used by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, La Tronche, France, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and regulatory constraints, and because no data-sharing plan is defined in the study protocol.

REFERENCES:
- [Background] Coste B, Houge G, Murray MF, Stitziel N, Bandell M, Giovanni MA, Philippakis A, Hoischen A, Riemer G, Steen U, Steen VM, Mathur J, Cox J, Lebo M, Rehm H, Weiss ST, Wood JN, Maas RL, Sunyaev SR, Patapoutian A. Gain-of-function mutations in the mechanically activated ion channel PIEZO2 cause a subtype of Distal Arthrogryposis. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):4667-72. doi: 10.1073/pnas.1221400110. Epub 2013 Mar 4. PMID 23487782
- [Background] Felsenthal N, Zelzer E. Mechanical regulation of musculoskeletal system development. Development. 2017 Dec 1;144(23):4271-4283. doi: 10.1242/dev.151266. PMID 29183940
- [Background] Nowlan NC. Biomechanics of foetal movement. Eur Cell Mater. 2015 Jan 2;29:1-21; discussion 21. doi: 10.22203/ecm.v029a01. PMID 25552425
- [Background] Pollard AS, McGonnell IM, Pitsillides AA. Mechanoadaptation of developing limbs: shaking a leg. J Anat. 2014 Jun;224(6):615-23. doi: 10.1111/joa.12171. Epub 2014 Mar 18. PMID 24635640
- [Background] Hoff JM, Loane M, Gilhus NE, Rasmussen S, Daltveit AK. Arthrogryposis multiplexa congenita: an epidemiologic study of nearly 9 million births in 24 EUROCAT registers. Eur J Obstet Gynecol Reprod Biol. 2011 Dec;159(2):347-50. doi: 10.1016/j.ejogrb.2011.09.027. Epub 2011 Oct 17. PMID 22005589
- [Background] Lowry RB, Sibbald B, Bedard T, Hall JG. Prevalence of multiple congenital contractures including arthrogryposis multiplex congenita in Alberta, Canada, and a strategy for classification and coding. Birth Defects Res A Clin Mol Teratol. 2010 Dec;88(12):1057-61. doi: 10.1002/bdra.20738. Epub 2010 Nov 15. PMID 21157886
- [Background] Darin N, Kimber E, Kroksmark AK, Tulinius M. Multiple congenital contractures: birth prevalence, etiology, and outcome. J Pediatr. 2002 Jan;140(1):61-7. doi: 10.1067/mpd.2002.121148. PMID 11815765
- [Background] Dahan-Oliel N, Cachecho S, Barnes D, Bedard T, Davison AM, Dieterich K, Donohoe M, Fafara A, Hamdy R, Hjartarson HT, S Hoffman N, Kimber E, Komolkin I, Lester R, Ponten E, van Bosse HJP, Hall JG. International multidisciplinary collaboration toward an annotated definition of arthrogryposis multiplex congenita. Am J Med Genet C Semin Med Genet. 2019 Sep;181(3):288-299. doi: 10.1002/ajmg.c.31721. Epub 2019 Jul 7. PMID 31282072